CLINICAL TRIAL: NCT07134777
Title: Mechanisms of Visual Restoration After Occipital Stroke (MOVROS)
Brief Title: Mechanisms of Visual Restoration After Occipital Stroke
Acronym: MOVROS
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Research to Prevent Blindness (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Mental Health (NIMH) (NIH); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Krystel Huxlin, Professor of Ophthalmology, University of Rochester
Other Study IDs: STUDY00010767; 1U01NS136338-01 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cortical Blindness; Stroke Ischemic; Vision Loss Partial; Visual Fields Hemianopsia; Hemianopia; Hemianopia Homonymous; Occipital Lobe Infarct
Keywords: occipital stroke; vision loss; Homonymous quadranopsia
MeSH Terms: conditions — Blindness, Cortical; Ischemic Stroke; Hemianopsia; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cortically Blind Subjects: Subjects must exhibit unilateral stroke or stroke-like damage to primary visual cortex or its immediate afferent white matter sustained within the specified age range of 21 - 80 years.
  Interventions: Diagnostic Test: MRI
- Control Subjects: Subjects with no history of neurological disorders and normal cognitive abilities.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Functional MRI scan

SUMMARY:
This project will collect brain imaging data to quantify the effects of early visual cortex damage and visual training interventions on the structure and function of the residual visual system. Our goal is to improve understanding of the consequences of permanent visual cortex damage in humans, and to understand how visual training impacts the function of the residual visual system to restore perception.

ELIGIBILITY:
Cortically Blind Subjects (n=50)

Inclusion:

* Subjects between 21 and 80 years of age
* Subjects must be residents of the United States or Canada
* Subjects must exhibit unilateral stroke or stroke-like damage to primary visual cortex or its immediate afferent white matter sustained within the specified age range of 21 - 80 years (verified by MRI and/or CT scans)
* Subjects with reliable visual field defects in both eyes (homonymous defects) as measured by Humphrey, MAIA, Goldmann, and/or equivalent perimetry. This deficit must be large enough to enclose a 5-deg diameter visual stimulus.
* Subjects must be able to fixate on visual targets reliably for 1000ms, with jitter over less than 1-deg of visual angle.

  o Note: This will be initially assessed by review of visual field reports as supplied by subjects during the screening process. However, we will be unable to fully assess their fixation ability until they start the psychophysics testing in our lab. If at that time we discover that they are unable to maintain adequate fixation, they will be withdrawn from the study.
* Subjects must be willing, able, and competent to provide their own informed consent
* Subjects must have their own home computer (desktop or laptop) and reliable internet access
* All subjects must have normal cognitive abilities and memory, sufficient to be able to understand and follow written and oral instructions in English, as well as to remember how to complete visual training at home, on their own, as instructed, for several months.
* Justification: We can only accept English-speaking subjects due to a lack of resources for supporting those who would require interpreter services. As all of our subjects are required to spend 3-5 days in lab with rigorous testing and training requirements, we must be able to communicate clearly and with minimal misunderstandings. This would require for up to 5-full days of in person interpreter services, for which we do not have funding. Additionally, ongoing communications take place by phone, email, and/or text as a part of home training (for routine check-ins and technical support for example) in the intervals between laboratory visits. This would require us to essentially have "on demand" access to interpreter services, which is simply not feasible.
* Subjects must be safe and willing to undergo magnetic resonance imaging (MRI) scans

Exclusion:

* Subjects who have past or present ocular disease interfering with visual acuity
* Subjects with best-corrected visual acuity (BCVA) worse than 20/40 in either eye
* Subjects who have documented or suspected damage to the dorsal Lateral Geniculate Nucleus
* Subjects who have diffuse whole-brain degenerative processes
* Subjects who have experienced traumatic brain injury
* Subjects who have any other brain damage deemed by study staff to potentially interfere with training ability or outcome measures
* Subjects who have oculomotor defects deemed by study staff to potentially interfere with training ability or outcome measures (i.e., by impairing stable fixation during testing or training)
* Subjects who have documented history of drug/alcohol abuse
* Subjects who are currently taking neuroactive medications which would impact training, as determined by PI
* Subjects who have cognitive, memory or seizure disorders
* Subjects with one-sided attentional neglect
* Subjects who lack the competence or are otherwise unable to perform the visual training exercises as directed.
* Subjects who have contradictions to MRI scanning will be excluded. These contraindications include: a) central nervous system aneurysm clips; b) implanted neural stimulator; c) implanted cardiac pacemaker or defibrillator; d) cochlear implant; e) ocular foreign body (e.g., metal shavings); f) insulin pump; g) metal shrapnel or bullet; h) any implanted device that is incompatible with MRI.
* Subjects who have conditions that preclude MRI scanning, e.g., morbid obesity, claustrophobia.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cortically blind patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Identify visual areas of damage | Baseline, Visit 2, Optional visits 3-7
  Use fMRI scans to identify areas of damage
Characterize visual response prior to visual training | Baseline, Visit 2, Optional visits 3-7
  Visual responses of different brain areas spared by the patients stroke will be analyzed using a population receptive field (pRF) method.
Characterize how visual response properties in residual visual areas change following a period of visual training | Baseline, Visit 2, Optional visits 3-7
  Characterize how visual response properties in residual visual areas change following a period of visual training. Visual responses of different brain areas will be analyzed using a population receptive field (pRF) method.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States